CLINICAL TRIAL: NCT00455832
Title: Influence of Ribavirin and Interferon on Semen Quality, IRIS Study
Acronym: IRIS
Status: Completed | Type: Observational
Sponsor: Foundation for Liver Research (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRIS Study
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-02

CONDITIONS: Sperm Motility (Focus of Study)
Keywords: sperm chromatin structure integrity; sperm concentration; sperm motility; sperm morphology; peginterferon; ribavirin; hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: peginterferon alpha and ribavirin — sperm collection

SUMMARY:
The aim of this study is to study the effect of peginterferon alpha and ribavirin on spermatozoa.

DETAILED DESCRIPTION:
During and six months after treatment with peginterferon alpha and ribavirin strict use of birth control is recommended (the producers advice two reliable forms) for both men and women because ribavirin has teratogenic and/or embryo-lethal effects in animal studies.

In cases of pregnancies during paternal exposure to peginterferon alpha and ribavirin elective termination of the pregnancy is usually recommended. However three cases of births after paternal exposure are reported with no birth defects. Cases of abnormalities after paternal exposure to ribavirin are lacking.

Also studies on the influence of ribavirin on sperm in human are lacking.

The aim of this study is to study the effect of peginterferon alpha and ribavirin on spermatozoa in men using these medication.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Treatment with peginterferon and ribavirin in the presence of a chronic Hepatitis C infection

Exclusion Criteria:

* Preexisting semen abnormalities.
* Concurrent use of drugs influencing sperm concentration,motility and morphology.
* Less then one million spermatozoa/ml in semen at screening.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2006-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J de Knegt, MD PhD, Principal Investigator — Foundation for Liver Research
Locations (1):
- Erasmus M C, University Medical Center Rotterdam, Rotterdam, Netherlands